CLINICAL TRIAL: NCT03953885
Title: Fire Needle Therapy on Plaque Psoriasis With Blood Stasis Syndrome: A Randomized, Single-blind, Multicentre Clinical Trial
Brief Title: Fire Needle Therapy on Plaque Psoriasis With Blood Stasis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shaanxi Provincial Hospital of Traditional Chinese Medicine (Unknown); The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other); Shijiazhuang Hospital of Traditional Chinese Medicine (Unknown); Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018YFC1705303-02
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Blood stasis syndrome; Randomized controlled trial; Fire Needle Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fire needle group (Experimental): Participants in experimental group will receive Fire needle therapy once a week for 4 weeks.In addition, participants will receive basic treatment, including the use of moisturizing lotion, avoid induction and aggravating factors, proper bathing to clean the skin, reasonable lifestyle and treatment.
  Interventions: Other: Fire needle
- Fire needle placebo group (Placebo Comparator): Participants in experimental group will receive Fire needle placebo therapy once a week for 4 weeks.In addition, participants will receive basic treatment, including the use of moisturizing lotion, avoid induction and aggravating factors, proper bathing to clean the skin, reasonable lifestyle and treatment.
  Interventions: Other: Fire needle Placebo

INTERVENTIONS:
Other: Fire needle — 1. Participants wear eye masks and fully expose the lesions. After selecting the acupuncture points, the surgeon routinely disinfects the hands of the operator and the acupuncture points of the participants before the operation. After selecting an acupuncture needle with a specification of 0.4*40mm and ignites the alcohol lamp, the operator continuously moves the needle from the needle root to the needle tip to burn the red needle to disinfect the needle in the outer flame of the alcohol lamp.
  2. The operator ignites the alcohol lamp, and burns the needle tip and the needle body to the outer flame of the alcohol lamp until it is completely red (the length of the needle burning red is determined by the acupuncture depth), and then rapidly penetrates the skin lesion vertically, the depth of the acupuncture is based on the thickness of the skin lesion, when the operation is performed, the outer edge of the lesion is punctured to the center point, and the spacing is 0.3 to 0.5 cm.
  Arms: Fire needle group
Other: Fire needle Placebo — 1. Participants wear eye masks and fully expose the lesions (no lesions on the head and face, external genitalia and skin folds). After selecting the acupuncture points, the surgeon routinely disinfects the hands of the operator and the acupuncture points of the participants before the operation, then selects an acupuncture needle with a specification of 0.4*40mm to prepare for operation.
  2. The operator rapidly penetrates the skin lesion vertically, the depth of the acupuncture is based on the thickness of the skin lesion, when the operation is performed, the outer edge of the lesion is punctured to the center point, and the spacing is 0.3 to 0.5 cm.
  Arms: Fire needle placebo group

SUMMARY:
This study was designed as a multicenter, randomized, single blinded and placebo-controlled clinical trial. The aim of the study is to evaluate the clinical efficacy, safety and control of recurrence rate of plaque psoriasis with blood stasis syndrome, after treated with fire needle therapy.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease characterized by the complex interaction between the immune system, related susceptibility loci, autoantigens and various environmental factors. In China, the prevalence is about 0.47%. Current treatment strategies for psoriasis mainly focus on developing new drugs that disrupt IL-23 or IL-17 cytokine, but this targeted therapy is not effective for all patients. A growing body of evidence indicates that psoriasis-related damage is not limited to the skin, but is closely related to coronary heart disease, stroke, metabolic syndrome, and chronic kidney disease. These comorbidities have, to a certain extent, increased mortality in patients with psoriasis. Traditional Chinese medicine (TCM) has always been used to treat patients with psoriasis in China. Blood stasis syndrome is one of the basic syndromes of psoriasis. which accumulates in meridians, viscera and limbs to form a variety of syndromes with psoriasis for a long time and is similar to many metabolic related diseases. Fire needle therapy is one of the traditional Chinese specialty treatments, which has effects of warming yang to expel cold, warming and activating meridian, dispersing stasis and relieving pain. Studies have shown that fire needle therapy of plaque psoriasis in stationary phase is effective, with fewer side effects, and can reduce the recurrence rate. This multicenter, randomized, single-blind, placebo-controlled trial will objectively and standardly evaluate the clinical effectiveness, safety and control of recurrence of fire needle therapy to obtain objective evidence of international standards and form clinical norms suitable for popularization and application.

ELIGIBILITY:
Inclusion Criteria:

1. Comply with the diagnostic criteria of Western medicine for plaque psoriasis and the diagnostic criteria for TCM syndromes;
2. Skin lesions involve ≤10% BSA (the lesions are mainly located in the trunk and/or limbs, palm/sole, face/scalp, vulva area is not included);
3. Age between 18 and 65 years old;
4. Those who voluntarily participate in the study and sign informed consent.

Exclusion Criteria:

1. Patients with erythrodermic, arthritic, pustular or punctate psoriasis;
2. Other active skin diseases may affect the condition assessment;
3. Received research drugs, biological agents and immunosuppressive agents within 1 month;
4. 2 weeks of treatment with topical glucocorticoids, phototherapy, etc.;
5. During severe, uncontrollable local or systemic acute or chronic infections;
6. Patients with severe systemic diseases; or clinical test indicators in one of the following conditions: alanine aminotransferase or aspartate aminotransferase increased by >1.5 times the upper limit of normal; creatinine increased by 1.5 times the upper limit of normal; blood routine indicators (white blood cell count) Any one of the red blood cell count, hemoglobin amount, and platelet count) is below the lower limit of normal; or other laboratory abnormalities are judged by the investigator to be unsuitable for participation in the trial;
7. A history of malignant tumors and patients with primary or secondary immunodeficiency and hypersensitivity;
8. Such surgery will be required during major surgery or study during 8 weeks;
9. Pregnant or lactating women;
10. A person with a history of alcohol abuse, drug abuse or drug abuse;
11. Have a history of serious mental illness or family history;
12. Other reasons researchers believe that it is inappropriate to participate in this research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis area and severity index (PASI) | Up to 56 days after treatment
  Psoriasis Area and Severity Index (PASI) involves grading psoriatic plaques based on erythema (E), infiltration (I), desquamation (D). Severity is graded from 0-4 for each criteria (0 - none, 1 - slight, 2 - moderate, 3 - severe, and 4 - very severe). The body is divided into 4 regions, head, upper extremities, trunk, and lower extremities, and for each region, the surface area involvement is graded on a 0-6 scale (0 - 0% involvement, 1 - <10%, 2 - 10-<30%, 3 - 30-<50%, 4 - 50-<70%, 5 - 70-<90%, 6 - 90-100%).The highest potential PASI score is 72, with higher PASI scores indicating worse psoriasis.

SECONDARY OUTCOMES:
Body surface area (BSA) | Up to 56 days after treatment
  The percentage of body surface area (BSA) involved in psoriasis is estimated by fingerprinting, where the entire palm of the patient represents approximately 1% of the total BSA. The number of handprints on psoriasis skin in a body part is used to determine the extent to which the body part is affected by psoriasis (%)
Physician Global Assessment (PGA) | Up to 56 days after treatment
  Physician Global Assessment (PGA) is scored on a 5-point scale, reflecting a global consideration of the erythema (E), infiltration (I), desquamation (D) across all psoriatic lesions. It is calculated as follows: PGA score = (E + I + D) / 3, then the score needs to be rounded to the nearest whole number [PGA scale: Clear (0) - Very Severe (5)].
Dermatology Life quality index(DLQI) | Up to 28 days after treatment
  The Dermatology Life Quality Index (DLQI) is a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores range from 0-30, a higher score indicating a greater impact on a participant's quality of life.
Patient-reported quality of life (PRQoL) | Up to 28 days after treatment
  Patient-reported quality of life (PRQoL) is used to assess the impact of psoriasis on individual social life. Scores range from 0-25, a higher score indicating a greater impact on a participant's social life.
Visual Analogue Score (VAS) | Up to 56 days after treatment
  Visual Analog Scale (VAS) is used to measure lesion pruritus from 0 to 100 mm at eash visit (with 0 being no pruritis and 100 being maximum pruritis).
TCM syndrome score | Up to 56 days after treatment
  The TCM symptom score is used to assess changes in blood syndrome related symptoms during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Department of dermatology, Shanghai Yueyang Integrated Medicine Hospital, Shanghai
Locations (5):
- China (5):
  - Shijiazhuang Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - First Affiliated Hospital of Heilongjiang Chinese Medicine University, Harbin, Heilongjiang
  - Affiliated hospital of jiangxi university of traditional Chinese medicine, Nanchang, Jiangxi
  - Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Hospital of Traditional Chinese Medicine, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu L, Lu Y, Yan XN, Yang SQ, Gong LP, Li LE, Zhao YD, Yin QF, Wang RP, An YP, Huang G, Zhang JF, Sun XY, Li X, Li B. Efficacy and safety of fire needle therapy for blood stasis syndrome of plaque psoriasis: protocol for a randomized, single-blind, multicenter clinical trial. Trials. 2020 Aug 25;21(1):739. doi: 10.1186/s13063-020-04691-7. PMID 32843084